CLINICAL TRIAL: NCT06388876
Title: The Effect of Exercise Interventions on Post-traumatic Stress Disorder and Sleep Quality in Young Individuals Directly Affected by the 2023 Kahramanmaraş Earthquakes in Türkiye: A Randomized Controlled Double-Blind Study
Brief Title: The Effect of Exercise on Post-traumatic Stress Disorder and Sleep Quality in Individuals Affected by the 2023 Kahramanmaraş Earthquakes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Bahar Anaforoglu, assoc.prof, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AnkaraYBUbk
Record Dates: First submitted 2024-04-22; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Earthquake; Stress Disorders, Post-Traumatic
Keywords: natural disaster; earthquake; exercise; post-traumatic stress disorder; sleep quality; physiotherapy and rehabilitation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Motor Activity; Sleep Initiation and Maintenance Disorders | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: there are 2 groups; exercise and control
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Exercise group did aerobic exercise during 6 weeks. Also this group took advice including lifestyle.
  Interventions: Other: Exercise; Other: lifestyle advice
- control (Experimental): Control group only took advice including lifestyle.
  Interventions: Other: lifestyle advice

INTERVENTIONS:
Other: Exercise — Members of the exercise group received an exercise intervention twice a week for six weeks accompanied by a physiotherapist.
  Other Names: lifestyle advice
  Arms: Exercise
Other: lifestyle advice — At the beginning of the program, the members of the individuals were given lifestyle recommendations, both verbally and in writing (in the form of a brochure) within the scope of a common training initiative.The individuals groups received both written (brochure) and verbal training within the scope of lifestyle recommendations (the effects of planned and regular exercise, sleep problems, methods of coping with stress, etc.).

SUMMARY:
Natural disasters can have adverse impacts on both physical and mental health. Post-traumatic stress disorder (PTSD) and sleep disorders are among the most common problems seen after natural disasters. Exercise may represent a safe, cost-effective, accessible, non-pharmacological method for treating PTSD and sleep problems. The aim of this study was to investigate the effect of exercise interventions on PTSD and sleep quality in young individuals affected by the 2023 Kahramanmaraş earthquakes in Türkiye.

ELIGIBILITY:
Inclusion Criteria:

* age 18-30
* being directly affected by the earthquake in Mardin
* providing voluntary consent to participating in the study

Exclusion Criteria:

* involvement in an existing active regular exercise program
* the presence a physical problem capable of preventing exercise
* the presence of severe psychiatric disorders or cognitive and/or perceptual problems
* regular use of sedative or neuropsychiatric drugs
* active alcohol or drug addiction
* missing assessment parameters
* failure to participate in the intervention programs, or not continuing wıth the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Post-traumatic Stress Disorder Short Scale | 6 weeks
  This self-report Likert-type scale was developed by LeBeau et al. in order to assess post-traumatic stress symptoms. The scale consists of nine questions and a single dimension. Each question is scored between 0 for "Not at all" and 4 for "Extremely". Total possible scores range between 0 and 36. The higher the total score, the higher the level of Post-traumatic Stress Disorder . The cut-off value of the scale was calculated as 24
Pittsburgh Sleep Quality Index | 6 weeks
  The Pittsburgh Sleep Quality Index consists of 24 questions and seven categories that yield information about the type and severity of sleep disturbance experienced in the past month. The Pittsburgh Sleep Quality Index includes questions assessing sleep quality, transition time, duration, efficiency, disturbance, sleep medication use, and daytime dysfunction due to sleep problems. Each item is scored from 0 (no distress at all) to 3 (severe distress). Total possible scores range from 0 to 21. A higher score means poorer sleep quality. A total score of 0-5 is regarded as indicating healthy sleep, 6-10 as poor sleep, and above 10 as long-term sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: bahar külünkoğlu, assoc. prof., Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yildirim Beyazıt University, Ankara, Turkey (Türkiye)